CLINICAL TRIAL: NCT02879058
Title: The Effect of Intraoperative Contact Sonography on Quality of Life Following Laparoscopic or Robotic Myomectomy
Brief Title: Intraoperative Ultrasound in Laparoscopic or Robotic Myomectomy Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to inadequate enrollment.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Katherine Smith, Clinical fellow, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLA- 16-031
Record Dates: First submitted 2016-07-25; First posted 2016-08-25 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Fibroid Uterus; Quality of Life
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without Ultrasound (No Intervention): Laparoscopic or robotic myomectomy will be performed without aid of intraoperative contact ultrasonography
- With Ultrasound (Experimental): Laparoscopic or robotic myomectomy will be performed with aid of intraoperative contact ultrasonography
  Interventions: Procedure: Intraoperative contact ultrasonography

INTERVENTIONS:
Procedure: Intraoperative contact ultrasonography — In patients randomized to myomectomy with contact ultrasonography, the laparoscopic or robotic ultrasound probe will be advanced through an existing port site into the pelvis after traditional myomectomy has been performed. The face of the ultrasound transducer will be guided over the uterus (including open hysterotomy sites) in systematic strokes, taking special care to note locations of myomas that may have been missed by the preceding excision. Additional hysterotomy sites will be made as necessary in order to remove persistent myomas. Any number of additional ultrasound passes and excisions may be performed in order to achieve the most comprehensive removal of myomas.
  Arms: With Ultrasound

SUMMARY:
This study evaluates whether use of intraoperative ultrasound during laparoscopic or robotic myomectomy impacts quality of life. Half of participants will undergo laparoscopic or robotic myomectomy with use of the intraoperative ultrasound and half will undergo traditional laparoscopic or robotic myomectomy.

DETAILED DESCRIPTION:
In full acknowledgement of the correlation between complete leiomyoma exeresis and symptom relief, the investigators hypothesize that use of contact ultrasonography at the time of laparoscopic or robotic myomectomy will enable improved identification and extraction of uterine fibroids which will, in turn, lead to a greater improvement in quality of life among those women who receive intraoperative ultrasound compared to those who do not. In this blinded randomized controlled trial, the investigators will augment traditional laparoscopic and robotic myomectomy with intraoperative ultrasound in half the symptomatic patients enrolled in the study. The other half will be randomized to undergo laparoscopic or robotic myomectomy without use of intra-operative ultrasound. Both groups will complete Uterine Fibroid Symptom and Quality of Life (UFS- QOL) questionnaires before and after surgery (6 months post procedure) to determine whether use of laparoscopic contact ultrasonography has a positive impact on patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal and nonpregnant
2. Advised to undergo laparoscopic or robotic myomectomy by their provider
3. Documented imaging with transvaginal ultrasound or pelvic MRI within the past year, which accurately and within reason documents the location and number of leiomyomas present within the uterus
4. If deemed necessary by the provider, must have a pelvic MRI prior to surgery that states there are no concerning findings for malignancy
5. Must be eligible to undergo laparoscopic surgery and willing to present for clinic and imaging follow up during the 6 months following myomectomy
6. Must understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Appearance of uterus concerning for malignancy on pelvic MRI
2. Current pregnancy
3. Any contraindication to laparoscopic or robotic surgery
4. Treatment with gonadotropin-releasing hormone (GnRH) analogs in the past 36 months

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Measured at baseline (before surgery) and 6 months post-surgery
  Symptom and health-related quality of life will be measured by The Uterine Fibroid Symptom and Quality of Life (UFS-QOL) questionnaire administered to all study participants before myomectomy and 6 months post-myomectomy.

SECONDARY OUTCOMES:
Operating Time | Measured at surgery
  Operating time is defined as the total period of time from when the procedure starts until the procedure is deemed complete.
Blood Loss | Measured at surgery
  Blood loss (in mL) will be estimated for all procedures by the primary surgeon and gleaned from the anesthesia operative flowsheet.
Weight of Excised Myomas | Measured at the time of Pathology evaluation.
  After extraction, all myomas will be submitted to pathology. Their cumulative weight will be measured by the Pathologist and gleaned by the research team from the final pathology report.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Zimberg, MD, Principal Investigator — Cleveland Clinic Florida; Katherine A Smith, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Selected de-identified ultrasound images and surgical data will be shared with BK Ultrasound, the manufacturer of the ultrasound device.

REFERENCES:
- [Background] Shimanuki H, Takeuchi H, Kikuchi I, Kumakiri J, Kinoshita K. Effectiveness of intraoperative ultrasound in reducing recurrent fibroids during laparoscopic myomectomy. J Reprod Med. 2006 Sep;51(9):683-8. PMID 17039695
- [Background] Nezhat FR, Roemisch M, Nezhat CH, Seidman DS, Nezhat CR. Recurrence rate after laparoscopic myomectomy. J Am Assoc Gynecol Laparosc. 1998 Aug;5(3):237-40. doi: 10.1016/s1074-3804(98)80025-x. PMID 9668143
- [Background] Mais V, Ajossa S, Guerriero S, Mascia M, Solla E, Melis GB. Laparoscopic versus abdominal myomectomy: a prospective, randomized trial to evaluate benefits in early outcome. Am J Obstet Gynecol. 1996 Feb;174(2):654-8. doi: 10.1016/s0002-9378(96)70445-3. PMID 8623802
- [Background] Radosa MP, Owsianowski Z, Mothes A, Weisheit A, Vorwergk J, Asskaryar FA, Camara O, Bernardi TS, Runnebaum IB. Long-term risk of fibroid recurrence after laparoscopic myomectomy. Eur J Obstet Gynecol Reprod Biol. 2014 Sep;180:35-9. doi: 10.1016/j.ejogrb.2014.05.029. Epub 2014 Jun 2. PMID 25016181
- [Background] Fedele L, Parazzini F, Luchini L, Mezzopane R, Tozzi L, Villa L. Recurrence of fibroids after myomectomy: a transvaginal ultrasonographic study. Hum Reprod. 1995 Jul;10(7):1795-6. doi: 10.1093/oxfordjournals.humrep.a136176. PMID 8582982
- [Background] Hanafi M. Predictors of leiomyoma recurrence after myomectomy. Obstet Gynecol. 2005 Apr;105(4):877-81. doi: 10.1097/01.AOG.0000156298.74317.62. PMID 15802421
- [Background] Fauconnier A, Chapron C, Babaki-Fard K, Dubuisson JB. Recurrence of leiomyomata after myomectomy. Hum Reprod Update. 2000 Nov-Dec;6(6):595-602. doi: 10.1093/humupd/6.6.595. PMID 11129693
- [Background] Doridot V, Dubuisson JB, Chapron C, Fauconnier A, Babaki-Fard K. Recurrence of leiomyomata after laparoscopic myomectomy. J Am Assoc Gynecol Laparosc. 2001 Nov;8(4):495-500. doi: 10.1016/s1074-3804(05)60610-x. PMID 11677326
- [Background] Piccolboni P, Settembre A, Angelini P, Esposito F, Palladino S, Corcione F. Laparoscopic ultrasound: a surgical "must" for second line intra-operative evaluation of pancreatic cancer resectability. G Chir. 2015 Jan-Feb;36(1):5-8. PMID 25827662
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Manyonda IT, Bratby M, Horst JS, Banu N, Gorti M, Belli AM. Uterine artery embolization versus myomectomy: impact on quality of life--results of the FUME (Fibroids of the Uterus: Myomectomy versus Embolization) Trial. Cardiovasc Intervent Radiol. 2012 Jun;35(3):530-6. doi: 10.1007/s00270-011-0228-5. Epub 2011 Jul 20. PMID 21773858
- [Background] Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92. doi: 10.1097/01.MLR.0000062554.74615.4C. PMID 12719681